CLINICAL TRIAL: NCT06546085
Title: Extracellular Vesicles, Insulin Action, and Exercise on Vascular Function in Type 2 Diabetes
Brief Title: Extracellular Vesicles, Insulin Action, and Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Virginia (Other)
Responsible Party: Principal Investigator, Steven K Malin, PhD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2024000230; R01DK133598-01A1 (NIH)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a between-within clinical trial study design. Groups (lean, obese/normal glucose tolerance, type 2 diabetes) will be matched on age and sex while those with obesity and normal glucose tolerance (NGT) will have matched BMI to type 2 diabetes (T2D) for cross-sectional comparisons. People with obesity and NGT as well as obesity with T2D will undergo exercise training for 16 weeks to determine EV changes in comparison to lean controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lean with Normal Glucose Tolerance (No Intervention): Participants will not receive the study intervention and will be healthy controls.
- Obesity with Normal Glucose Tolerance (Experimental): Participants with obesity and normal glucose tolerance will participate in 3 supervised exercise training sessions at 85% VO2max that expends ~400 kcal for 16 weeks.
  Interventions: Behavioral: Exercise
- Obesity with Type 2 Diabetes (Experimental): Participants with obesity and type 2 diabetes will participate in 3 supervised exercise training sessions at 85% VO2max that expends ~400 kcal for 16 weeks.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Supervised treadmill exercise at 85% VO2max, 3x/wk for 16 weeks. Exercise duration will be adjusted based on individual VO2-heart rate (HR) relationship so that ~400 kcals will be expended during each training session.
  Arms: Obesity with Normal Glucose Tolerance; Obesity with Type 2 Diabetes

SUMMARY:
Extracellular vesicles (EVs) play a role in obesity-induced insulin resistance and likely impact the development of cardiovascular disease. However, little is known on how EVs affect vascular insulin action in people. The purpose of this study is to understand how EVs play a role in type 2 diabetes related cardiovascular disease. This research will also study if exercise can change how EVs impact blood flow and metabolic health. This study will contribute to designing precision medicine to treat/prevent cardiovascular disease in type 2 diabetes.

DETAILED DESCRIPTION:
Insulin resistance is a key underlying factor promoting hyperglycemia and hypertension in people with type 2 diabetes (T2D), who have a 3-fold greater cardiovascular disease (CVD) risk when compared with healthy controls. Despite several therapeutic approaches that favor insulin sensitivity through a variety of purported mechanisms (e.g. weight loss, incretins, AMPK activation, reduction in bioactive lipids: DAG/ceramides, etc.), long-term progression of glucose deterioration occurs. This suggests adjunctive targets may be important to prevent/reverse T2D. Studies show that extracellular vesicles (EVs) obtained from plasma are involved in obesity-induced insulin resistance at levels of adipocytes, muscle, and liver. However, little is known how plasma EVs affect vascular insulin action in humans. This is of clinical relevance as EVs enhance the Framingham Risk Score, suggesting EVs are a unique factor promoting CVD. This proposal will fill this knowledge gap by conducting a translational study in 3 distinct groups of people separated by obesity and T2D. The investigators hypothesize that 1) insulin will promote EV uptake and modify insulin signaling in endothelial cells, 2) EVs from adults with T2D will impair vessel reactivity compared to controls; 3) insulin will alter circulating EV insulin signaling and cargo, and 4) exercise training will change EV uptake and cargo as well as EV mediated vascular reactivity to insulin as well as relate to improved vascular function in humans.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 30 - 80 years old.
* HbA1c <5.7% and fasting glucose <100mg/dl to be considered NGT
* T2D diagnosis or confirmation HbA1c ≥6.5% and fasting glucose ≥126 mg/dl
* Prescribed metformin, GLP-1 agonists (oral/injectable), TZDs, DPP-IV inhibitors, Acarbose, SGLT-2 inhibitors ≥6 year.
* Has a body mass index of 20-24.99 or 25.0-45 kg/m2.
* Not diagnosed with Type 1 diabetes.
* Not currently engaged in >150 min/wk of exercise.

Exclusion Criteria:

* Participants with morbid obesity (BMI >45 kg/m2) and underweight patients (BMI: ≤18 kg/m2).
* Intolerance to insulin
* Evidence of type 1 diabetes and diabetics requiring insulin therapy.
* Participants who have not been weight stable (≥2 kg weight change in past 6 months)
* Participants who have been recently active in past 6 months via health screening questions (≥150 min of moderate/high intensity exercise)
* T2D with HbA1c ≥10.0%
* Participants who are smokers or who have quit smoking ≤2 years ago
* Participants prescribed metformin, GLP-1 agonists (oral/injectable), TZDs, DPP-IV inhibitors, Acarbose, SGLT-2 inhibitors within 6 year.
* Hypertriglyceridemic (≥400 mg/dl) and hypercholesterolemic (≥260 mg/dl) participants as determined from LabCorp samples.
* Kidney dysfunction as determined from LabCorp biochemical outcomes (e.g. creatinine (≥1.0 mg/dl), eGFR (≤59 ml/min/1.73), BUN (≥24 mg/dl) as derived from comprehensive metabolic panels).
* Hypertensive (≥160/100 mmHg) at time of screening.
* Abnormal liver function (reflective from comprehensive panel liver enzymes Alk (≥121 IU/L), AST (≥40 IU/L) and ALT (≥32 IU/L) via LabCorp).
* History of significant metabolic, cardiac, cerebrovascular, hematological, pulmonary, gastrointestinal, liver, renal, or endocrine disease or cancer that in the investigator's opinion would interfere with or alter the outcome measures, or impact subject safety.
* Pregnant (as evidenced by positive pregnancy test) or nursing women
* Participants with contraindications to participation in an exercise training program
* Known hypersensitivity to perflutren (contained in Definity).
* Anemic as confirmed by hematocrit (HCT) (women ≤36%, Men ≤38%) at time of screening.
* Suggested infections at time of screening as confirmed by WBC (≥10.8 x10E3/uL) and/or platelets (≥450 x10E3/uL).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Change in Extracellular Vesicles during insulin infusion | From enrollment to the end of treatment at 16 weeks.
  Extracellular vesicles (CD41 -CD31+, CD45, Tx, CD31, CD105) will be isolated from plasma before and during insulin stimulation.

SECONDARY OUTCOMES:
Change in Metabolic Insulin Sensitivity by the Isoglycemic Clamp | From enrollment to the end of treatment at 16 weeks.
  Measure of glucose metabolism determined by the glucose infusion during the last 30 minutes of the 150 clamp procedure.
Change in Contrast Enhanced Ultrasound | From enrollment to the end of treatment at 16 weeks.
  Measure of microvascular blood flow before and during insulin stimulation.
Change in Flow Mediated Dilation of the brachial artery | From enrollment to the end of treatment at 16 weeks.
  Measure of blood flow using ultrasound before and during insulin stimulation.
Change in Pulse Wave Velocity | From enrollment to the end of treatment at 16 weeks.
  Measure of arterial stiffness using pulse waves at the carotid and femoral arteries before and during insulin stimulation.
Change in Augmentation Index | From enrollment to the end of treatment at 16 weeks.
  Measure of aortic pressure waveforms before and during insulin stimulation.
Change in Post Ischemic Flow Velocity in the brachial artery | From enrollment to the end of treatment at 16 weeks.
  Measure of blood flow using ultrasound before and during insulin stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Malin, PhD, Principal Investigator — Rutgers University - New Brunswick
Locations (3):
- United States (3):
  - Institute for Food, Nutrition, and Health, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Clinical Research Center, New Brunswick, New Jersey
  - Rutgers University Loree Gymnasium, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang M, Wang L, Chen Z. Research progress of extracellular vesicles in type 2 diabetes and its complications. Diabet Med. 2022 Sep;39(9):e14865. doi: 10.1111/dme.14865. Epub 2022 May 20. PMID 35509124
- [Background] Nozaki T, Sugiyama S, Koga H, Sugamura K, Ohba K, Matsuzawa Y, Sumida H, Matsui K, Jinnouchi H, Ogawa H. Significance of a multiple biomarkers strategy including endothelial dysfunction to improve risk stratification for cardiovascular events in patients at high risk for coronary heart disease. J Am Coll Cardiol. 2009 Aug 11;54(7):601-8. doi: 10.1016/j.jacc.2009.05.022. PMID 19660689
- [Background] Ragland TJ, Heiston EM, Ballantyne A, Stewart NR, La Salvia S, Musante L, Luse MA, Isakson BE, Erdbrugger U, Malin SK. Extracellular vesicles and insulin-mediated vascular function in metabolic syndrome. Physiol Rep. 2023 Jan;11(1):e15530. doi: 10.14814/phy2.15530. PMID 36597186
- [Background] Heiston EM, Ballantyne A, Stewart NR, La Salvia S, Musante L, Lanningan J, Erdbrugger U, Malin SK. Insulin infusion decreases medium-sized extracellular vesicles in adults with metabolic syndrome. Am J Physiol Endocrinol Metab. 2022 Oct 1;323(4):E378-E388. doi: 10.1152/ajpendo.00022.2022. Epub 2022 Jul 20. PMID 35858245
- [Background] Heiston EM, Ballantyne A, La Salvia S, Musante L, Erdbrugger U, Malin SK. Acute exercise decreases insulin-stimulated extracellular vesicles in conjunction with augmentation index in adults with obesity. J Physiol. 2023 Nov;601(22):5033-5050. doi: 10.1113/JP282274. Epub 2022 Feb 16. PMID 35081660
- [Background] Eichner NZM, Gilbertson NM, Heiston EM, Musante L, LA Salvia S, Weltman A, Erdbrugger U, Malin SK. Interval Exercise Lowers Circulating CD105 Extracellular Vesicles in Prediabetes. Med Sci Sports Exerc. 2020 Mar;52(3):729-735. doi: 10.1249/MSS.0000000000002185. PMID 31609300
- [Background] Hallmark R, Patrie JT, Liu Z, Gaesser GA, Barrett EJ, Weltman A. The effect of exercise intensity on endothelial function in physically inactive lean and obese adults. PLoS One. 2014 Jan 20;9(1):e85450. doi: 10.1371/journal.pone.0085450. eCollection 2014. PMID 24465565
- [Background] Steinberg HO, Chaker H, Leaming R, Johnson A, Brechtel G, Baron AD. Obesity/insulin resistance is associated with endothelial dysfunction. Implications for the syndrome of insulin resistance. J Clin Invest. 1996 Jun 1;97(11):2601-10. doi: 10.1172/JCI118709. PMID 8647954
- [Background] Solomon TP, Malin SK, Karstoft K, Haus JM, Kirwan JP. The influence of hyperglycemia on the therapeutic effect of exercise on glycemic control in patients with type 2 diabetes mellitus. JAMA Intern Med. 2013 Oct 28;173(19):1834-6. doi: 10.1001/jamainternmed.2013.7783. No abstract available. PMID 23817567